CLINICAL TRIAL: NCT00025142
Title: A Study of ZD1839 (Iressa) in Combination With Oxaliplatin, 5-Fluorouracil (5-FU) and Leucovorin (LV) in Advanced Solid Malignancies (Phase I) and Advanced Colorectal Cancers (Phase II)
Brief Title: Gefitinib and Combination Chemotherapy in Treating Patients With Advanced Solid Tumors or Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: SUMC-670; CDR0000068923 (Registry Identifier: PDQ (Physician Data Query)); NCI-4370
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2005-02

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Fluorouracil; Gefitinib; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: gefitinib
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Biological therapies such as gefitinib may interfere with the growth of tumor cells and slow the growth of the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug with gefitinib may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of gefitinib and oxaliplatin combined with leucovorin and fluorouracil in treating patients who have advanced solid tumors or colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of gefitinib and oxaliplatin when combined with fluorouracil and leucovorin calcium in patients with advanced solid tumors. (Phase I) (Phase I closed as of 5/30/02)
* Determine the pharmacokinetics and pharmacodynamics of this regimen in these patients.
* Determine the dose-limiting toxic effects and other toxic effects of this regimen in these patients.
* Determine the antitumor response in patients with advanced colorectal adenocarcinoma treated with this regimen. (Phase II)
* Determine the overall survival and time to progression in patients with advanced colorectal adenocarcinoma treated with this regimen. (Phase II)
* Determine the presence of polymorphisms or other genetic alterations in genes implicated in the action of this regimen and determine their possible relationship with toxic effects of and antitumor response to this regimen in these patients.

OUTLINE: This is a dose-escalation study of gefitinib and oxaliplatin (L-OHP).

* Phase I (closed as of 5/30/02): Patients receive L-OHP IV over 2 hours on day 1 and leucovorin calcium (CF) IV over 2 hours followed by fluorouracil (5-FU) IV bolus and 5-FU IV over 22 hours on days 1 and 2 during all courses. Beginning with course 2, patients also receive oral gefitinib daily on days 1-14. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response (CR) receive 2 additional courses past CR.

Sequential dose escalation of gefitinib is followed by sequential dose escalation of L-OHP. Cohorts of 3-6 patients receive escalating doses of gefitinib and L-OHP until the maximum tolerated dose (MTD) of the combination is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients are stratified according to prior therapy:

  * Stratum A: Received no prior therapy or received adjuvant 5-FU/CF or adjuvant 5-FU/CF/irinotecan at least 6 months ago
  * Stratum B: Received prior therapy for metastatic disease or received adjuvant 5-FU/CF fewer than 6 months ago or prior irinotecan Patients receive therapy as in phase I (closed as of 5/30/02) with L-OHP and gefitinib at the recommended phase II dose.

PROJECTED ACCRUAL: Approximately 12-15 patients will be accrued for phase I of the study within 4-6 months (Phase I closed as of 5/30/02). A total of 30-81 patients (18-46 for stratum A and 12-35 for stratum B) will be accrued for phase II of the study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Phase I (closed as of 5/30/02):

  * Histologically confirmed metastatic or unresectable solid tumor for which standard curative or palliative measures do not exist or are no longer effective
* Phase II:

  * Histologically confirmed metastatic or unresectable colorectal adenocarcinoma
* Measurable disease or assessable but nonmeasurable disease (including ascites, pleural/pericardial effusions, lymphangitis cutis/pulmonis, inflammatory breast disease, abdominal masses (not followed by CT scan/MRI), or cystic lesions)

  * Disease characterized only by elevated serum tumor marker allowed
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy:

* More than 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm ^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST/ALT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No ongoing or active infection
* No peripheral neuropathy
* No prior allergic reactions to compounds of similar chemical or biologic composition to gefitinib or other study agents
* No other concurrent uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior bone marrow or stem cell support with high-dose chemotherapy
* At least 24 hours since prior colony-stimulating growth factors

Chemotherapy:

* See Biologic therapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No more than 3 prior chemotherapy regimens

Endocrine therapy:

* At least 2 weeks since prior hormonal therapy except megestrol for anorexia/cachexia

Radiotherapy:

* No prior pelvic or whole abdominal radiotherapy
* At least 4 weeks since other prior radiotherapy and recovered

Surgery:

* At least 4 weeks since prior major surgery (e.g., laparotomy) and recovered

Other:

* At least 4 weeks since prior investigational therapy
* No other concurrent investigational or commercial anticancer agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-07; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Branimir I. Sikic, MD, Study Chair — Stanford University
Locations (1):
- Stanford Cancer Center at Stanford University Medical Center, Stanford, California, United States

REFERENCES:
- [Result] Fisher GA, Kuo T, Ramsey M, Schwartz E, Rouse RV, Cho CD, Halsey J, Sikic BI. A phase II study of gefitinib, 5-fluorouracil, leucovorin, and oxaliplatin in previously untreated patients with metastatic colorectal cancer. Clin Cancer Res. 2008 Nov 1;14(21):7074-9. doi: 10.1158/1078-0432.CCR-08-1014. PMID 18981005
- [Result] Kuo T, Cho CD, Halsey J, Wakelee HA, Advani RH, Ford JM, Fisher GA, Sikic BI. Phase II study of gefitinib, fluorouracil, leucovorin, and oxaliplatin therapy in previously treated patients with metastatic colorectal cancer. J Clin Oncol. 2005 Aug 20;23(24):5613-9. doi: 10.1200/JCO.2005.08.359. PMID 16110021
- [Result] Cho CD, Fisher GA, Halsey JZ, et al.: A phase I study of ZD1839 (Iressa) in combination with oxaliplatin, 5-fluorouracil (5-FU) and leucovorin (LV) in advanced solid malignancies. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-38, 2002.